CLINICAL TRIAL: NCT03096002
Title: Small Steps for Big Changes: A Lifestyle Program to Reduce the Risk of Developing Type 2 Diabetes in the Community
Brief Title: Small Steps for Big Changes: A Lifestyle Program to Reduce the Risk of Developing Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mary Jung, Assistant Professor, University of British Columbia
Other Study IDs: H16-02028
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: PreDiabetes
Keywords: PreDiabetes, Lifestyle intervention, Exercise Behavior, Adherence
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lifestyle change (one-treatment group): The lifestyle change program is a 3-week program that will introduce participants to a regular healthy lifestyle that includes exercising at least three times per week and the program will highlight simple dietary strategies. There is no randomization to this program - all individuals enrolled will partake in the same program and will be followed up for 12 months after the program has concluded.
  Interventions: Behavioral: Lifestyle change

INTERVENTIONS:
Behavioral: Lifestyle change — The 3-week lifestyle change program will introduce participants to a regular healthy lifestyle including exercise and dietary changes for reducing sugar intake, reducing refined/processed carbohydrate intake, increasing vegetable consumption. The 3-week program will include six supervised exercise sessions and three exercise sessions performed independently (e.g., at home or outside of the lab). The supervised session will include brief behavioral counseling sessions that teach participants self-regulatory skills to promote independence and long-term adherence to exercising and dietary changes.

SUMMARY:
The purpose of this study is to address whether inactive individuals with prediabetes who take part in the Small Steps for Big Changes program, which is a 3-week supervised exercise and lifestyle change program with brief counseling, will be more adherent to regular exercise one year after program completion compared to before they took part in the program.

DETAILED DESCRIPTION:
The study is a one-group repeated measures design and the primary outcome is exercise adherence at 12 months post the 3-week supervised exercise program. There is no randomization of individuals to conditions. Exercise adherence will be measured using self-report physical activity (using the Godin leisure time exercise questionnaire) and a subsample will also wear tri-axial accelerometers to measure total time spent in moderate-to-vigorous physical activity assessed over 7 days. Secondary outcomes include physical fitness, haemoglobin A1C, quality of life, self-regulatory efficacy, anthropometrics, diet and exercise-related cognitive errors.

The 3-week lifestyle program includes six sessions with a lifestyle coach and exercise sessions performed at home. These sessions will focus on regular healthy lifestyle that includes walking (or exercise of any kind) at least three times per week and will highlight simple dietary strategies that are linked to reduced risk of T2D. The 3-week supervised exercise program includes brief exercise counseling sessions that teach participants self-regulatory skills to promote independence and long-term adherence to exercise and a healthy diet. At the conclusion of the three-week program, participants will be asked to continue exercising a minimum of three times per week for twelve months on their own.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak and read English
* BMI between 25-40 kg/m2 (as measured by body mass and height self-reporting),
* blood pressure of <160/99 mm Hg assessed according to CHEP guidelines,
* not diagnosed with type 2 diabetes
* no prior history of cardiovascular disease
* not on hormone replacement therapy
* Cardiovascular medications (e.g., statins) will be allowed if the participant is on stable therapy (6 months on same dose).

Exclusion Criteria, if subjects:

* take glucose-lowering medications that have changed within the past 6 months;
* report any explicit contraindications to exercise (e.g., musculoskeletal injury, chest pain during exercise)
* report having had a heart attack or stroke in the past;
* report that they are pregnant or plan on becoming pregnant over the next 12 months;
* have uncontrolled major depression;
* have bone or joint problem (for example, back, knee, or hip) that could be made worse by a change in physical activity which a physician has not cleared them for to exercise;
* report that a physician has not cleared their participant for exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit a community-based sample of adults living with prediabetes.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
minutes of moderate to vigorous physical activity | change from before participants begin the program to 52 weeks after they finish the program for 7 consecutive days
  objective measure of physical activity will be measured using tri-axial accelerometers in a subsample of ~100 participants
independent bouts of physical activity | change from when participants begin the program to 52 weeks after they finish the program
  self-reported measure of bouts of physical activity as assessed by the Godin Leisure Time Exercise Questionnaire

SECONDARY OUTCOMES:
glucose control | change from when participants begin the program to 52 weeks after they finish the program (week 55)
  haemoglobin A1C
Aerobic fitness | before the program begins (week 0), after the program is completed (week 3), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  six-minute walk test
Perceived health-related quality-of-life | before the program begins (week 0), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  SF-12 Health Survey (Ware, Kosinski, & Keller, 1995)
Self-regulatory efficacy for physical activity and diet | before the program begins (week 0), after the program is completed (week 3), 4-weeks after the completion of the program (week 7), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  questionnaire
minutes of moderate to vigorous physical activity | 24 weeks after program completion (week 27) for 7 consecutive days
  objective measure of physical activity will be measured using tri-axial accelerometers in a subsample of ~100 participants
independent bouts of physical activity | 4- (week 7) and 24-weeks (week 27) after completion of the program
  self-reported measure of bouts of physical activity as assessed by the Godin Leisure Time Exercise Questionnaire

OTHER OUTCOMES:
blood pressure | before the program begins (week 0), after the program is completed (week 3), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  mean arterial blood pressure assessed manually
weight | before the program begins (week 0), after the program is completed (week 3), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  body weight assessed by objective scale
waist circumference | before the program begins (week 0), after the program is completed (week 3), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  circumference of the waist assessed manually
reach | before the program begins (week 0)
  reach of the program as assessed by RE-AIM
dietary adherence | before the program begins (week 0), 24 weeks after completion of the program (week 27), and 52 weeks after completion of the program (week 55)
  brief food frequency questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- YMCA of Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No